CLINICAL TRIAL: NCT00941746
Title: A Randomised, Double-blind, Placebo-controlled, Single Ascending Dose, Phase I Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of PG110 (Anti-NGF Monoclonal Antibody) in Patients With Pain Attributed to Osteoarthritis of the Knee
Brief Title: Safety and Tolerability of PG110 in Patients With Knee Osteoarthritis Pain
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Jerry A Hall, Medical Director, Abbott
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: PG110-01; 2008-006219-19 (EudraCT Number)
Record Dates: First submitted 2009-07-14; First posted 2009-07-20 (Estimated); Last update posted 2011-06-07 (Estimated); Status verified 2011-05

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (9):
- Lowest dose of PG110 (Experimental): single, slow intravenous infusion
  Interventions: Biological: PG110
- Second dose of PG110 (Experimental): single, slow intravenous infusion
  Interventions: Biological: PG110
- Third dose of PG110 (Experimental): single, slow intravenous infusion
  Interventions: Biological: PG110
- Fourth dose of PG110 (Experimental): single, slow intravenous infusion
  Interventions: Biological: PG110
- Fifth dose of PG110 (Experimental): single, slow intravenous infusion
  Interventions: Biological: PG110
- Top dose of PG110 (Experimental): single, slow intravenous infusion
  Interventions: Biological: PG110
- Placebo (Experimental): single, slow intravenous infusion that matches PG110 in appearance
  Interventions: Biological: Placebo
- Seventh Dose of PG110 (Experimental): single, slow intravenous infusion
  Interventions: Biological: PG110
- Eight Dose of PG110 (Experimental): single, slow intravenous infusion
  Interventions: Biological: PG110

INTERVENTIONS:
Biological: PG110 — Single, slow intravenous infusion
  Arms: Lowest dose of PG110
Biological: PG110 — Single, slow intravenous infusion
  Arms: Second dose of PG110
Biological: PG110 — Single, slow intravenous infusion
  Arms: Third dose of PG110
Biological: PG110 — Single, slow intravenous infusion
  Arms: Fourth dose of PG110
Biological: PG110 — Single, slow intravenous infusion
  Arms: Fifth dose of PG110
Biological: PG110 — Single, slow intravenous infusion
  Arms: Top dose of PG110
Biological: PG110 — Single, slow intravenous infusion
  Arms: Seventh Dose of PG110
Biological: PG110 — Single, slow intravenous infusion
  Arms: Eight Dose of PG110
Biological: Placebo — Single, slow intravenous infusion that matches PG110 in appearance
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of a single intravenous dose of PG110, a monoclonal antibody that inhibits the effects of the naturally occurring substance, nerve growth factor (NGF).

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe pain attributed to knee osteoarthritis

Exclusion Criteria:

* Significant comorbidity
* Significant pain states other than osteoarthritis
* Concomitant medications that might affect assessments

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2009-08; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
The number and severity of adverse events | Three months

SECONDARY OUTCOMES:
Terminal elimination half-life | Three months
Dose proportionality of the area under the serum concentration-time curve | Three months
Pain in the index knee | Three months
Western Ontario and McMaster Universities questionnaire | Three months

CONTACTS AND LOCATIONS:
Overall Officials: Jerry Hall, MD, Study Director — Abbott
Locations (1):
- Site Ref # / Investigator 51568, Utrecht, Netherlands